CLINICAL TRIAL: NCT05644691
Title: Impact of the Daily Use of the Tested Emollient on Corticosteroids Consumption in Patients Minimum 3 Years Old With Atopic Dermatitis (SCORAD 20-30) Versus Their Usual Emollient
Brief Title: Impact of the Daily Use of Emollient on Corticosteroids Consumption in Patients With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP19002-LIPIKAR BAUME AP+M
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; corticosteroids; SCORAD
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lipikar Baume AP+M: The group applies Lipikar Baume AP+M twice daily for 3 months. Participants have 4 visits (Day0, Day 28, Day56, Day84) with different outcome measures including self-evaluations).
  Interventions: Other: Lipikar Baume AP+M
- Usual emollient: The group applies their usual emollient twice daily for 3 months. Participants have 4 visits (Day0, Day28, Day56, Day84 with different outcome measures including self-evaluations).
  Interventions: Other: Usual emollient

INTERVENTIONS:
Other: Lipikar Baume AP+M — application of Lipikar Baume AP+M twice daily for 3 months in parallel with the corticosteroid treatment
  Groups: Lipikar Baume AP+M
Other: Usual emollient — application of the usual emollient twice daily for 3 months in parallel with the corticosteroid treatment
  Groups: Usual emollient

SUMMARY:
This study aims at assessing the reduction of consumption of corticosteroids (same mid-potent corticosteroids for all patients) afforded by the use of a specific emollient in comparison to the usual one in subjects suffering from atopic dermatitis.

DETAILED DESCRIPTION:
The study is conducted in compliance, as closely as possible, with the current version of the world medical association declaration of Helsinki, local regulations based on International Council on Harmonisation (ICH) guidelines for Good Clinical Practice.

The primary objective of this study is to compare the tested emollient and the usual emollient through the weight of used dermocorticosteroid. The weight of used dermocorticosteroid is compared at the end of the study by a Student t-test (or a non parametric Wilcoxon test depending on the data distribution).

The following hypotheses are used for the estimation of the sample size calculation:

* Power (1 - β) = 80%
* Two-sided significance level (α) = 5%
* Expected inter-group difference = 0.6g
* Standard deviation = 1.4g.

Statistical analyses is performed with SAS® version 9.4 or higher (SAS institute, North Carolina, USA).

Continuous variables are summarized as number of observations, mean, standard deviation, standard error, median, minimum and maximum (95% confidence interval will be provided if necessary). For categorical variables, subject counts and percentages will be provided.

Analyses use 2-sided tests at the 5% significance level, except the normality tested at the threshold of 1% (Shapiro-Wilk test).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of atopic dermatitis must meet Hanifin's criteria (at least 3 basic features and at least 3 minor features)
* mild atopic dermatitis present for at least 6 months before inclusion (SCORAD at inclusion between 20 and 30)
* able to apply the emollient (each morning and evening) during a three-month period

Exclusion Criteria:

* presenting with another dermatological condition that could interfere with clinical evaluation
* having received any systemic treatment, including PUVAtherapy for atopic dermatitis in the month prior to Day 0
* who intend to expose themselves to the sun during the trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients meeting the inclusion and exclusion criteria and agreeing to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
efficacy of treatments | from baseline to Day84
  the efficacy of treatments is evaluated by corticosteroids consumption (weight of product and number of applications)

SECONDARY OUTCOMES:
change in SCORing Atopic Dermatitis (SCORAD) measure | from baseline to Day84
  evaluation of SCORAD by the dermatologist in relation with the emollient consumption (weight of product and number of applications)
change in Patient-Oriented SCORing Atopic Dermatitis (PO-SCORAD) measure | from baseline to Day84
  evaluation of PO-SCORAD by the patient in relation with the emollient consumption (weight of product and number of applications)
change in LOCAL SCORing Atopic Dermatitis (LOCAL SCORAD) measure | from baseline to Day84
  evaluation of LOCAL SCORAD by the dermatologist in relation with the emollient consumption (weight of product and number of applications)
change in cutaneous discomfort | from baseline to Day84
  evaluation of skin sensation (itching, tingling, burning) by the patient on a 4-point scale (from absence to severe)
change in global efficacy | from Day28 to Day84
  evaluation of global efficacy by the patient on a 4-point scale (from nil to excellent)
change in global tolerance | from Day28 to Day84
  evaluation of global tolerance of the treatment (emollient + corticosteroid) by the patient on a 4-point scale (from nil to excellent)
change in Patient Benefit Index (PBI) measure | from baseline to Day84
  questionnaire filled in by the patient or the patient's parents (whether the statement applies to the situation or not, possible answers: not at all, somewhat, moderately, quite, very, does not apply to me)
change in the quality of life (patients aged 18 years or over) | from baseline to Day84
  questionnaire about the Atopic Burden Scale for Adults (ABS-A) with the following scale: never, rarely, sometimes, often, very often, constantly, not applicable. A higher score means a higher burden.
change in the quality of life (patients aged less than 18 years) | from baseline to Day84
  questionnaire about the Atopic Dermatitis Burden Scale for the Family (ABS-F) with the following scale: no, without hesitation; I don't know; maybe; yes, without hesitation; not applicable. A higher score means a higher burden.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Le Floc'h, Study Director — Cosmetique Active International
Locations (1):
- DOST, Svidník, Slovakia